CLINICAL TRIAL: NCT06680700
Title: Controlled Desaturation Study for Perin Health Patch Pulse Oximetry Validation
Brief Title: Controlled Desaturation Study for Perin Health Patch Validation
Status: Recruiting | Type: Observational
Sponsor: Perin Health Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: PHD-004-24
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Oxygen Saturation Measurement
Keywords: Pulse Oximeter; Oxygen Saturation; Wearable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy adult volunteers aged 18-50, who meet strict inclusion criteria to ensure safety and consistency in the results. Participants must be in good general health, with no history of respiratory, cardiovascular, or other systemic diseases that could pose additional risks during controlled desaturation. All participants are fully vaccinated for COVID-19, fluent in English, and capable of understanding and complying with the study procedures.
  Interventions: Device: Perin Health Patch

INTERVENTIONS:
Device: Perin Health Patch — The Perin Health Patch (PHP) is a non-invasive, chest-worn device designed to monitor blood oxygen saturation (SpO2) and additional vital signs, including heart rate, respiratory rate, ECG, and bioimpedance (BioZ). Unlike traditional fingertip pulse oximeters, the PHP integrates multi-wavelength photoplethysmography (PPG) sensors with ECG and BioZ technology, allowing for continuous SpO2 tracking even during movement and daily activities.

SUMMARY:
This study aims to test the accuracy of the Perin Health Patch (PHP), a non-invasive, chest-worn device that measures blood oxygen levels, by comparing its readings to a standard pulse oximeter device. The PHP device uses light sensors to measure blood oxygen saturation (SpO2), similar to how standard pulse oximeters work, and could allow for continuous remote monitoring at home. Participants in this study will breathe low-oxygen air through a mask to simulate different oxygen levels in a controlled environment. The goal is to see if the PHP device can accurately measure blood oxygen levels under different conditions and meet safety standards set by the FDA and international guidelines.

DETAILED DESCRIPTION:
The Perin Health Patch (PHP) is a non-invasive, chest-worn medical device that continuously measures blood oxygen saturation (SpO2), alongside other vital signs. The PHP's performance will be assessed under controlled hypoxemia (low oxygen levels), where its readings will be compared to a standard pulse oximeter validated against co-oximeter reference values.

In this single-site, prospective study, up to 25 healthy adult volunteers will undergo controlled desaturation sessions. During each session, a mask delivering a low-oxygen gas mixture will be used to safely lower participants' SpO2 levels. This method simulates a range of oxygenation states, from 70% to 100% SpO2, which is critical for testing the device's accuracy across a clinically relevant range. The PHP's readings will be captured alongside those from two standard pulse oximeters placed on both hands. Participants will be carefully monitored by clinical staff throughout the study, with emergency oxygen and other medical equipment readily available to ensure participant safety.

Participants will complete two desaturation "runs," each lasting approximately 10-15 minutes, with brief breaks between sessions. During some sessions, participants may be asked to walk slowly on a treadmill to simulate movement conditions. This study design aligns with the ISO 80601-2-61 standard, supporting robust accuracy assessments under both stationary and motion conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years to 50 years
* The subject is in good general health with no evidence of any medical problems,
* Fully vaccinated for COVID-19
* Fluent in both written and spoken English
* Willing and able to provide informed consent,
* Able to comply with study procedure.

Exclusion Criteria:

* Children (under the age of 18)
* Adults above 50 years old
* History of heart, lung, kidney, or liver disease.
* Obesity (BMI > 30),
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Diagnosis of Raynaud's disease
* Unacceptable collateral circulation based on an exam by the investigator (Allen's test).
* Pregnant, lactating or trying to get pregnant
* Current smoker
* History of diabetes
* Clotting disorder
* Hemoglobinopathy or history of anemia
* History of fainting or vasovagal response
* Any other serious systemic illness
* Any other condition which, in the opinion of the investigators, would make them unsuitable for the study,
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly,
* Any evidence, in the opinion of the investigators, of medical problems or poor general health
* Any symptoms related to COVID-19
* No vaccinated for COVID-19
* Recent injection with methylene blue
* History of reactions to medical adhesives,
* Unable or unwilling to provide informed consent,
* Inability to comply with the study procedure,
* Non-English Speaker.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy adult volunteers recruited from the general community surrounding Woodland Hills, CA. The population is selected to ensure a controlled environment with minimal health variability, allowing for a precise assessment of the Perin Health Patch's performance in measuring blood oxygen saturation (SpO2) and other physiological metrics under controlled conditions of hypoxemia. All participants will be screened for general health and suitability to participate in a desaturation study, ensuring a homogenous, low-risk sample for accurate device validation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of SpO2 Measurements by Perin Health Patch Compared to Reference Pulse Oximeter | Immediately after the intervention
  The primary outcome measure is the accuracy of blood oxygen saturation (SpO2) readings from the Perin Health Patch (PHP) in comparison to those from a reference pulse oximeter. Accuracy will be determined by calculating the mean difference (bias) and standard deviation of differences (precision) between the SpO2 measurements obtained from the PHP and those from the reference devices across a range of hypoxemic conditions (70-100% SpO2).
  The PHP's SpO2 accuracy will be assessed using a root-mean-square difference (ARMS) in accordance with ISO 80601-2-61 standards, with a target ARMS of ≤ 4.0% SpO2 across the specified range.

SECONDARY OUTCOMES:
SpO2 Accuracy During Motion | Immediately after the intervention
  This outcome measures the accuracy of SpO2 readings from the PHP compared to a reference pulse oximeter while participants are in motion (e.g., walking on a treadmill). It specifically assesses if movement impacts the PHP's ability to maintain SpO2 accuracy within ISO 80601-2-61 standards, with a target ARMS of ≤ 4.0% SpO2.

CONTACTS AND LOCATIONS:
Overall Officials: Ian M McLane, Ph.D., Principal Investigator — Perin Health Devices
Locations (1):
- Perin Health Devices, Woodland Hills, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD), including de-identified datasets and a data dictionary describing collected variables, will be made available to other researchers following the completion of the study. The data will be shared in a way that maintains participant confidentiality and complies with ethical and legal standards. Access to IPD will be granted upon reasonable request and for use in research that aligns with the aims of the original study. Requests for IPD should be directed to the Principal Investigator, and access will be provided through a secure data-sharing platform after an approval process.
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT06680700/ICF_000.pdf